CLINICAL TRIAL: NCT04544254
Title: Effectivity of Bilateral Transversus Thoracis Muscle Plane Block to Reduce Pain and Stress Response After Open Heart Surgery: A Study to Interleukin-6 and Cortisol Plasma Concentration, Total Opioid Dose, and Time to First Opioid
Brief Title: Effectivity of Bilateral Transversus Thoracis Muscle Plane Block After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes056
Record Dates: First submitted 2020-08-29; First posted 2020-09-10 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Interleukin-6; Cortisol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral transversus thoracis muscle plane block (Active Comparator): Regional block will be performed after induction of anesthesia by anesthesiologist on duty who is not part of investigators for this study. The block will be performed in between intercostal space 4 and 5, lateral from sternum, with ultrasound guided
  Interventions: Procedure: Bilateral transversus thoracis muscle plane block
- Control (Placebo Comparator): Needle will be put in the superficial skin on the same area as transversus thoracis muscle plane block area without any drugs injected into the injection area
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Bilateral transversus thoracis muscle plane block — The block will be performed in between intercostal space 4 and 5, lateral from sternum, with ultrasound guided. Twenty milliliters bupivacaine 0.5% 1mg/body weight will be injected between internal intercostal muscle and transversus thoracis muscle on both sides.
  Arms: Bilateral transversus thoracis muscle plane block
Procedure: Control — A needle will be place in the similar area to the transversus thoracis muscle plane block, but no drugs will be injected to the area
  Arms: Control

SUMMARY:
This Study aimed to assess The Effectivity of Bilateral Transversus Thoracis Muscle Plane Block to Reduce Pain and Stress Response After Open Heart Surgery

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial. Thirty-two subject will be recruited with non-probability consecutive sampling method. Subjects who meet all inclusion criteria and do not have exclusion criteria will be asked to sign the informed consent form before included in this study. Subjects will be randomized into two groups. The first group is the treatment group who will get Bilateral Transversus Thoracis Muscle Plane Block after induction of anesthesia and the second group will be the control group who will not get any regional block during surgery. After surgery, time to first morphine dose, total morphine consumption in 24 hours, extubation time, and adverse events will be recorded for both group.

ELIGIBILITY:
Inclusion criteria:

1. Age 19-75 years old
2. Patients who will undergo elective open heart surgery with median sternotomy approach

Exclusion criteria:

1. Patient who does not agree to be included in this study
2. weight <45kg or >75 kg
3. Patient with chronic obstructive pulmonary disease
4. Patient with chronic kidney disease who needs regular hemodialysis.
5. Patient with local infection in the injection area for transversus thoracis muscle plane block
6. Patient with chronic pain
7. Patient with history of chronic analgetics drugs usage
8. Patient who is contraindicated for local anesthetics
9. Patient with communication disability
10. Patient with cognitive disorders
11. Patient with severe psychiatrics disorders, such as schizophrenia and bipolar disorder

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 plasma concentration | 48 hours
  Interleukin-6 plasma concentration will be measured 3 times, before surgery, 24 hours after surgery, and 48 hours after surgery
Cortisol plasma concentration | 48 hours
  cortisol plasma concentration will be measured 3 times, before surgery, 24 hours after surgery, and 48 hours after surgery

SECONDARY OUTCOMES:
total morphine dose | 24 hours
  investigators will record total morphine dose needed in 24 hours
time to first morphine | 24 hours
  investigators will record time to first morphine dose after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National General Hospital Dr. Cipto Mangunkusumo, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raksamani K, Wongkornrat W, Siriboon P, Pantisawat N. Pain management after cardiac surgery: are we underestimating post sternotomy pain? J Med Assoc Thai. 2013 Jul;96(7):824-8. PMID 24319854
- [Background] Roca J, Valero R, Gomar C. Pain locations in the postoperative period after cardiac surgery: Chronology of pain and response to treatment. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):391-400. doi: 10.1016/j.redar.2017.01.002. Epub 2017 Feb 22. English, Spanish. PMID 28237371
- [Background] Mello LC, Rosatti SF, Hortense P. Assessment of pain during rest and during activities in the postoperative period of cardiac surgery. Rev Lat Am Enfermagem. 2014 Jan-Feb;22(1):136-43. doi: 10.1590/0104-1169.3115.2391. PMID 24553714
- [Background] Li X, Feng Y, Yang BX. Postoperative pain after cardiac surgery. J Cardiothorac Vasc Anesth. 2010 Dec;24(6):1025-6. doi: 10.1053/j.jvca.2010.01.009. Epub 2010 Apr 22. No abstract available. PMID 20417122
- [Background] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] Jellish WS, Oftadeh M. Enhanced Recovery After Surgery for Cardiac Surgery: Will We Have the Techniques Needed to Reduce Opioid Use and Still Provide Appropriate Analgesia? J Cardiothorac Vasc Anesth. 2019 Feb;33(2):547-548. doi: 10.1053/j.jvca.2018.10.022. Epub 2018 Oct 24. No abstract available. PMID 30477887
- [Background] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Derived] Jaya AAGPS, Tantri AR, Heriwardito A, Mansjoer A. Single-centre, double-blind, randomised, parallel-group, superiority study to evaluate the effectiveness of general anaesthesia and ultrasound-guided transversus thoracis muscle plane block combination in adult cardiac surgery for reducing the surgical stress response: clinical trial protocol. BMJ Open. 2021 Nov 11;11(11):e051008. doi: 10.1136/bmjopen-2021-051008. PMID 34764171